CLINICAL TRIAL: NCT03111667
Title: A Hybrid Effectiveness-Implementation Trial of a School-Based Teen Marijuana Checkup
Acronym: TMCU5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Denise Walker, Research Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000988
Record Dates: First submitted 2017-03-20; First posted 2017-04-13 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Cannabis Use
Keywords: Marijuana; Motivational Enhancement Therapy; Adolescents
MeSH Terms: conditions — Marijuana Abuse | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Student Participants will be assigned in a 2:1 ratio to the Experimental "Teen Marijuana Check Up" or a Control "Treatment as Usual" condition.
  Interventionist Participants will be assigned in a 1:1 ratio to "Gold Standard" or "As Needed" Coaching
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Student Participants: Teen Marijuana Check Up (Experimental): 2 Session Motivational Enhancement Therapy intervention for adolescents who use marijuana.
  Interventions: Behavioral: Teen Marijuana Check Up
- Student Participants: Treatment As Usual (Other): Students will receive referrals to local agencies and other resources as typically done by school based staff. At the end of research follow-up period, students in this condition will be eligible to receive the active intervention.
  Interventions: Other: Treatment as Usual
- Interventionist Participants: Gold Standard Coaching (Experimental): Interventionists will receive weekly coaching and feedback about sessions and skills from the project PI.
  Interventions: Behavioral: Gold Standard Coaching
- Interventionist Participants: As Needed Coaching (Active Comparator): Interventionists will receive coaching and feedback about sessions and skills from the project PI only when sessions fall below adherent skill levels.
  Interventions: Behavioral: As Needed Coaching
- Administrator Participants: Environment (No Intervention): School Administrators will provide data about the school environment.
- School Staff Participants: Environment (No Intervention): Staff will provide data about the school environment

INTERVENTIONS:
Behavioral: Teen Marijuana Check Up — Two session Motivational Enhancement Therapy intervention. The first MET session relies on the use of motivational interviewing skills to hear the student's history and current concerns with marijuana. The second session involves the provision of a personalized feedback report based on the student's baseline assessment that reviews normative feedback on marijuana use, consequences experienced, money spent on marijuana, other drug and alcohol use, social supports for quitting and life goals.
  Arms: Student Participants: Teen Marijuana Check Up
Other: Treatment as Usual — Referral to community resources
  Arms: Student Participants: Treatment As Usual
Behavioral: Gold Standard Coaching — Weekly coaching and feedback about adherence to Motivational Interviewing Skills and intervention delivery in a group setting.
  Arms: Interventionist Participants: Gold Standard Coaching
Behavioral: As Needed Coaching — As needed coaching and feedback about adherence to Motivational Interviewing Skills and intervention delivery in an individual setting.
  Arms: Interventionist Participants: As Needed Coaching

SUMMARY:
A hybrid effectiveness-implementation trial that is designed to assess the effectiveness of an intervention (The Teen Marijuana Check-Up) when delivered in real world settings. In addition, the study will assess the frequency of coaching support needed by providers to maintain adherent skill levels.

DETAILED DESCRIPTION:
The objectives of the proposed study are to advance Type 2 translational science through an effectiveness-implementation "type 2" hybrid design to evaluate the clinical and cost-effectiveness of an efficacious intervention (Teen Marijuana Check-Up, TMCU) and compare the feasibility, acceptability, impact and cost-effectiveness of two integrity monitoring support systems. Marijuana continues to be the most frequently used drug in the U.S. and adolescent use is associated with negative effects such as academic failure, dropout, and emotional problems. Although marijuana is the most common presenting substance for 12-17 year olds seeking substance abuse treatment, few voluntarily seek indicated services. The TMCU is a brief, school-based motivational enhancement therapy approach that has been systematically evaluated in three randomized controlled trials with reliable beneficial effects in prompting voluntary participation in the intervention and decreasing adolescent marijuana use. With TMCU now well-positioned for broad dissemination, its public health impact may be enhanced by further research addressing: 1) to what extent its documented efficacy under controlled conditions translates to real-world effectiveness, and 2) what support systems are most useful in promoting sustained integrity in its delivery by the available school-based personnel. The proposed type 2 effectiveness/implementation hybrid trial will include randomization at multiple levels. Students will be randomly-assigned in a 1:2 ratio to 'services-as-usual' and TMCU intervention conditions, and school-based personnel identified to deliver TMCU will be randomly-assigned to do so under governance of a 'gold-standard' training/oversight support system (i.e., rapid, continual performance-based feedback and weekly coaching about integrity of TMCU delivery) or a less resource-intensive support system similarly including performance-based feedback but with process benchmarking (defined by prior performance of research interventionists in TMCU efficacy trials) prompting points at which these school-based personnel receive purveyor coaching. Expected trial participation of ten schools will enable recruitment of 30 TMCU interventionists, and access to a pool of 250 marijuana-using students during a two-year implementation period. This nested design (e.g., students in schools/intervention conditions; interventionists in schools/training/oversight support systems) will utilize multilevel models in study analyses to account for possible school-level clustering. A cost analysis will also be conducted. Longitudinal outcome and process data will be collected from school based staff (6, 12, 18, & 24 month follow-ups) and students (3 and 6 month followups).

The trial will occur in Washington state at an opportune time when legislative, fiscal, and socio-cultural factors converge to heighten potential adolescent exposure to marijuana-related harms-represents an effort by this investigative team to respond to such local challenges in a manner that will advance understanding of best practices for dissemination and implementation of this and other efficacious, school-based interventions

ELIGIBILITY:
Group 1: Administrators from local High Schools.

Inclusion Criteria:

* age 21 and older
* in an administrative role at one of the 10 participating high schools.

Exclusion Criteria:

* none

Group 2: School Staff- Climate Survey Respondents.

Inclusion Criteria:

* age 21 and older
* in a staff position at one of the 10 participating high schools.

Exclusion Criteria:

* none

Group 3: School Based Staff - Interventionists.

Inclusion Criteria:

* willing to participate in TMCU implementation procedures (i.e., randomization to coaching group, training, supervision and feedback, monitored performance via audio-recorded sessions),
* willing to share some personal demographic data,
* permission from supervisor,
* a two -year commitment and availability to participate in the project, and
* willingness to have sessions audio-recorded for feedback.

Exclusion Criteria: Otherwise eligible SBS will be excluded if

* plan to leave the school within the next year or,
* have an extended absence (e.g., 3 month parental leave, semester sabbatical) planned.

Group 4: Marijuana Using Students.

Inclusion Criteria:

* age (14-21 years old),
* grade (9-12)
* marijuana use
* willing to have sessions audio-recorded.

Exclusion Criteria: Individuals otherwise eligible will be excluded if:

* not fluent in English,
* have a thought disorder that precludes full participation, or
* refuse to accept randomization to condition.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Student Participants: Change in Number of Marijuana Use Days | baseline, 3, and 6 month follow-up
  self-reported, retrospective number of marijuana use days in the past 60.
School Based Interventionists - change in behavioral fidelity | within two weeks before training, 2 week, 6, 12, 18, and 24 month follow-up post training
  Adherent MITI score.

SECONDARY OUTCOMES:
School Based Interventionists - implementation acceptability | within two weeks before training, 2 week, 6, 12, 18, and 24 month follow-up post training
  School Based Interventionists - self-reported satisfaction with their experience in TMCU
Student Participants - change in marijuana related problems | baseline, 3, and 6 month follow-up
  self-reported retrospective marijuana problems

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Hartzler, PhD, Principal Investigator — University of Washington; Denise Walker, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Innovative Programs Research Group, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hartzler B, Lyon AR, Walker DD, Matthews L, King KM, McCollister KE. Implementing the teen marijuana check-up in schools-a study protocol. Implement Sci. 2017 Aug 10;12(1):103. doi: 10.1186/s13012-017-0633-5. PMID 28797270